CLINICAL TRIAL: NCT05114876
Title: Redesigning the Surgical Pathway: Optimizing PReOperative assessMent in Anesthesia Clinic for adulT Surgical Patients (PROMoTE)
Brief Title: Redesigning the Surgical Pathway (PROMoTE)
Acronym: PROMoTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5086
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Delirium; Cognitive Impairment; Perioperative/Postoperative Complications; Cognitive Dysfunction; Cognitive Decline
Keywords: perioperative neurocognitive disorders; postoperative delirium; delirium; pre-existing cognitive impairment
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Postoperative Complications; Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care
- Intervention (Active Comparator): Multicomponent delirium-risk prevention bundle
  Interventions: Other: Multicomponent delirium-risk prevention bundle

INTERVENTIONS:
Other: Multicomponent delirium-risk prevention bundle — This multidisciplinary intervention will introduce new practices including:
  1. Direct-to-Patient Education Program
  2. Directly informing anesthesia and surgery teams about high-risk patients by flagging their chart, and providing suggestions for POD mitigation
  3. Flag charts as high risk for POD so that nursing staff in both the PACU and the wards are aware, facilitating implementation of CHASM interventions (i.e. evidence-based delirium prevention protocols).
  4. Reinforce CHASM best practices with regular educational sessions for nurses.
  Arms: Intervention

SUMMARY:
Cognitive complications, that is problems with thinking and memory, are incredibly common after surgery, occurring in 10-50% of all older surgical patients. These complications can take different forms, but one of the most common is postoperative delirium (POD), a short-term state of confusion. In addition to being stressful for patients and their families, POD is linked to longer hospital stays, increased costs, higher mortality rates and other problems after surgery. Despite this, POD is often not recognized by doctors and there are currently no effective medications to treat POD. However, simple strategies such as helping patients to sleep properly and remain hydrated, have been shown to help.

This study is testing if a delirium-reduction program will reduce postoperative delirium (POD) in older surgical patients. The investigators will first test memory and thought processes before surgery to find people who are most likely to develop POD. Once these people have been identified, they will be enrolled in a program which includes recommendations for their care team (e.g. surgeon, anesthesiologist, nurses) as well as educational materials for them and their family related to things that can be done to prevent delirium. By identifying at-risk patients and making sure that their doctors and caregivers are aware of how to prevent delirium, the investigators expect that this study will make surgery safer for older surgical patients.

DETAILED DESCRIPTION:
Postoperative delirium (POD), an acute, reversible disturbance in brain function characterized by fluctuating levels of consciousness, attention and cognition is a common postoperative complication in older surgical patients. POD is associated with increased morbidity, mortality, and risk of dementia; in addition to longer hospital stays and increased healthcare costs. Despite this, POD frequently goes unrecognized by healthcare providers and is often poorly proactively managed. There are currently no effective pharmacological treatments for POD, although non-pharmacological prevention strategies (e.g. promoting sleep hygiene, hydration, and early mobilization) have proven effective.

This will be a two-phase, prospective, observational comparative study in patients (age ≥60) presenting for major, elective surgical procedures with an expected postoperative stay ≥1 day(s). In both phases, baseline cognitive screening will be used to identify individuals with evidence of pre-existing cognitive impairment (pre-CI), a key risk factor for POD, and only individuals with pre-CI will be eligible to continue in the study.

Phase I will establish the prevalence of POD and pre-CI in our patient population at Sunnybrook Health Sciences Centre, a tertiary care academic health sciences centre, and act as a control group for Phase II. Phase II will evaluate the effects of a comprehensive delirium-risk prevention bundle, which includes direct-to-patient education and healthcare provider awareness strategies. Participants in both Phase I and Phase II will provide written/verbal informed consent.

In each phase the study team will complete delirium assessments for 130 patients at baseline and on postoperative days 1-3. Demographic and clinical data will be abstracted from participants medical records. PHQ-9 (depression) and AD-8 (dementia screening interview) questionnaires will be completed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years old
* Undergoing major elective surgery (e.g., intra-abdominal, retroperitoneal, major orthopedic) with an expected postoperative stay of at least 1 night
* Evidence of cognitive impairment on baseline screening tests (i.e. any score < 90 on CBB or >10 on S-OMCT)

Exclusion Criteria:

* Patients undergoing cardiac surgery
* Patients undergoing intracranial neurosurgery
* Patients with known substance use disorder (verbally declared by patients)
* Unlikely to comply with study assessment (e.g., no fixed address, without access to internet/computer/phone).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of POD before and after implementation of an institutional prospective diagnostic program. | twice daily on postoperative days 1-3, morning/late afternoon
  POD evaluated by 3D-CAM and retrospectively using the CHART-DEL method

SECONDARY OUTCOMES:
Delirium Severity | twice daily on postoperative days 1-3, morning/late afternoon
  Assessed using CAM-S
Hospital length of stay | Until discharge, average of 1 week
  Duration of hospital admission in days
Unit adherence rate to CHASM principles | Until discharge, average of 1 week
  Unit adherence rate to CHASM principles

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participants data collected during this trial that underlie the results reported in the publication(s) will be available upon request after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon request immediately after publication of the primary results. No end date.
Access Criteria: Direct request to PI. Anyone who wishes to access the data.